CLINICAL TRIAL: NCT01456117
Title: A Phase 1, Multiple-Dose, Single-Blind Parallel Design, Single-Center, Dose-Ranging Study to Assess the Effects of Daily Administration of Pioglitazone for 14 Days on the Brain Hemodynamics of Healthy Elderly Subjects
Brief Title: Study to Assess the Effects of Daily Administration of Pioglitazone on Brain Hemodynamics in Healthy Elderly Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AD-4833/TOMM40_102; U1111-1125-0985 (Registry Identifier: WHO)
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: Drug Therapy; pharmacodynamics; pharmacokinetics
MeSH Terms: interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pioglitazone (Dose 1) QD (Experimental)
  Interventions: Drug: Pioglitazone
- Pioglitazone (Dose 2) QD (Experimental)
  Interventions: Drug: Pioglitazone
- Pioglitazone (Dose 3) QD (Experimental)
  Interventions: Drug: Pioglitazone
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone once daily for up to 14 days.
  Other Names: AD-4833; ACTOS
  Arms: Pioglitazone (Dose 1) QD
Drug: Pioglitazone — Pioglitazone once daily for up to 14 days.
  Other Names: AD-4833; ACTOS
  Arms: Pioglitazone (Dose 2) QD
Drug: Pioglitazone — Pioglitazone once daily for up to 14 days.
  Other Names: AD-4833; ACTOS
  Arms: Pioglitazone (Dose 3) QD
Drug: Placebo — Pioglitazone matching placebo once daily for up to 14 days.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to assess the effects of pioglitazone, once daily (QD), on brain hemodynamics in healthy elderly participants.

DETAILED DESCRIPTION:
The study will evaluate the effects on resting-state networks before and after therapeutic intervention, and also on task-related brain networks after specific cognitive challenges.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. The participant is a healthy adult male or female participant between the ages of 55 and 83 years, inclusive, at the time of informed consent and first dose of study medication dose.
4. Female participants of childbearing potential will not be included in the study. Female participants must be post-menopausal (defined as >2 years without menses).
5. The participant is considered to have normal cognitive abilities, as assessed by standard cognitive tests administered at the Screening visit. All participants will undergo a brief neuropsychological assessment which includes the Montreal Cognitive Assessment (MoCA) and Alzheimer Disease Cooperative Study Cognitive Function Screening Instrument to verify general cognitive status. Memory will be assessed with the Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Word List Memory Test and Trail Making Part B. Normal performance will be defined as scores within 1 standard deviation (SD) of age and education normative mean.

Exclusion Criteria:

1. The participant has received pioglitazone or any thiazolidinedione (TZD) in a previous clinical study or as a therapeutic agent within 1 year of Screening.
2. The participant is an immediate family member, study site employee (defined as study personnel and employees directly supervised by study personnel), or in a dependant relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
3. The participant has uncontrolled, clinically significant neurologic (e.g., migraines not well controlled, narcolepsy, previous head injury with loss of consciousness, or seizures), osteoporosis, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality which may impact the ability of the participant to participate or potentially confound the study results.
4. Participant has a known hypersensitivity or allergies to any component of the formulation of pioglitazone or related compounds.
5. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study. Participant is unwilling to agree to abstain from alcohol 24 hours prior to MRI or unwilling to abstain from drugs throughout the study.
6. History or evidence of any other central nervous system disorder that could be interpreted as a cause of dementia.
7. Current diagnosis of significant psychiatric disorders according to Diagnostic and Statistical Manual of Mental Disorders Forth Edition Text Revision (DSM-IV-TR). Subjects with recent/past psychiatric disorders who are currently in remission/asymptomatic without the use of medication may be eligible as determined by the principal investigator and the medical monitor.
8. Diabetes mellitus where the participant is being treated with insulin and/or peroxisome proliferator-activated receptor-ɣ (PPARɣ) agonist.
9. Participant has a history of cancer that required chemotherapy treatment within the past 2 years prior to Day 1, metastatic cancer in the past 5 years prior to Day 1, or radiation treatment to the brain in their lifetime. Subjects with basal cell or stage I squamous cell carcinoma of the skin will be eligible. Eligibility of subjects with a history of cancer will be determined by the principal investigator and medical monitor.10. History of macular edema, degeneration or any maculopathy.

11. Participant with a glycosylated hemoglobin (HbA1c) ≥6%. 12. Participant with congestive heart failure or significant edema (2+) of the extremities.

13. History of postmenopausal bone fracture (females only). 14. If male, the participant intends to donate sperm during the course of this study or for 30 days after the last dose of study drug.

15. Participant has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (i.e., a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn, or any surgical intervention [e.g., cholecystectomy]).

16. Participant has a positive test result for hepatitis B surface antigen (HBsAg), or hepatitis C antibody (anti-HCV) at Screening or a known history of human immunodeficiency virus infection (HIV).

17. Participant has a Screening or Check-in (Day 1) abnormal (clinically significant) ECG. (Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature by principal investigator. (If principal investigator is not a MD, ECG must be assessed by a qualified investigator).

18. Participant has abnormal Screening or Day 1 laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: Alanine Aminotransferase (ALT) and/or Aspartate Aminotransferase (AST) >2x the upper limits of normal (ULN).

19. Participant has a contraindication to having MRI, for example because of ferromagnetic foreign bodies (e.g., unremovable ferromagnetic dental work), medical devices such as aneurysm clips or cardiac pacemakers, or lead-based tattoos.

20. Participant has hematuria (microscopic or macroscopic) at Screening.

Ages: 55 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in BOLD fMRI Signal Related to Pioglitazone in Regions of the Brain Related to Cognition. | Baseline, Day 7 and Day 14.
  Regions of the brain related to cognition include the hippocampus and the dorsolateral prefrontal cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Clinical Science, Study Director — Takeda
Locations (1):
- Durham, North Carolina, United States